CLINICAL TRIAL: NCT05216562
Title: Efficacy and Safety of EXOSOME-MSC (Mesenchymal Stem Cell-Derived Exosomes) Therapy to Reduce Hyper-inflammation In Moderate COVID-19 (2019- New Corona Virus Disease) Patients
Brief Title: Efficacy and Safety of EXOSOME-MSC Therapy to Reduce Hyper-inflammation In Moderate COVID-19 Patients
Acronym: EXOMSC-COV19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dermama Bioteknologi Laboratorium (Industry)
Collaborators: Kementerian Riset dan Teknologi / Badan Riset dan Inovasi Nasional, Indonesia (Other Government)
Responsible Party: Principal Investigator, Bambang Darwono, Senior Clinical Consultant, Dermama Bioteknologi Laboratorium
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DBL-EXO-MSC-COV-19-CT-01; PPUK-RG.01.06.1.2.03.21.29 (Other: National Agency of Drug and Food Control of Indonesia)
Record Dates: First submitted 2022-01-28; First posted 2022-01-31 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: SARS-CoV2 Infection
Keywords: Mesenchymal Stemcells - derived Exosomes; SARS-COV-2, COVID-19; Hyper-inflammation; Cytokine Storm
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Group participants who receive injection of EXOSOME-MSC as adjuvant
  Interventions: Drug: Exosome-MSC Intravenous injection; Drug: COVID-19 Standard Treatment
- Control group (Placebo Comparator): Group participants who receive injection of Placebo (NaCL) as adjuvant
  Interventions: Drug: Placebo Intravenous Injection; Drug: COVID-19 Standard Treatment

INTERVENTIONS:
Drug: Exosome-MSC Intravenous injection — Intravenous injection of Exosome-MSC
  Other Names: Dermama Exosome-MSC
  Arms: Intervention group
Drug: Placebo Intravenous Injection — Intravenous injection of Placebo
  Other Names: Placebo
  Arms: Control group
Drug: COVID-19 Standard Treatment — Specific drugs considered standard treatment for COVID-10 by each location may vary
  Other Names: Drugs accepted as cures for COVID-19

SUMMARY:
In COVID-19 infection caused by the Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), there is a dysregulation of the immune system response that causes cytokine storm syndrome. SARS-CoV-2 works like a hijacker (hackers), sabotaging communication between cells so that the immune system, like T-cells, kills not only infected cells but also healthy cells. This dysregulation results in hyper-inflammation which cause damage to organs, not just the lungs. This is the cause of the high mortality rate in COVID-19 patients.

Exosomes are vesicles with a size of 30-100 nanometers originating from within cells that function to communicate with other cells. Exosomes are transport containers that contain bioactive cargo: such as proteins, genetic material, and various other molecules. These containers move from cells of origin, flowing through blood vessels or other body fluids to target cells. Exosomes penetrate the cell membrane and act on various organelles within the target cell.

All cell types can produce exosomes. What differentiates them is the cargo they contain. The exosome produced by mesenchymal stem cells (MSCs) contains bioactive cargo derived from mesenchymal stem cells, such as anti-inflammatory cytokines, growth factors, messengerRNA (mRNA) and microRNA (miRNA). The target cells are immune system cells, infected cells and progenitor cells from infected organs. On target immune cells, the anti-inflammatory cytokines work as immunomodulators to relieve hyper-inflammation. In infected cells, the miRNAs work to prevent viral replication by inhibiting the expression of SARS-CoV-2 virus RNA (viral mRNA silencing and degrading). In lung progenitor cells and other infected organs, the growth factors work to stimulate protein synthesis processes that function for organ regeneration.

This study is a multi-center, double-blind, randomized controlled trial (RCT) clinical trial with two arms: one intervention arm, and one control arm. The EXOSOME-MSC will be tested as adjuvant, on top of standard COVID-19 drugs. It will be injected to participants via intravenous route twice, in day-1 and day-7 of 14 days of study participation.

DETAILED DESCRIPTION:
The current study is a multi-center, double arm, adjuvant, randomized control trial (RCT), double-blind clinical trial, to analyze the differences in the usefulness and safety of Exosome-MSC intravenous injection therapy in moderate-grade COVID-19 patients with hyper-inflammation (Evans S.R, 2010).

This study used 2 groups (double arm) of study participants:

Treatment Group (Intervention Arm): received treatment in the form of standard therapy and injection of Exosomes-MSC.

Control Group (Control Arm): received treatment in the form of standard therapy and injection placebo.

The time interval for the implementation of the study protocol was 14 days. For each group (Treatment and Control) the minimum target number of participating patients and according to the inclusion criteria in this study were 30 people. The minimum total number of participants with 2 groups (Treatment and Control) is 60 people. (Rohrig B., 2010)

Random sample selection was carried out nationally from patients who entered the treatment room with a positive diagnosis of COVID-19 at the three Multi-Center Research Implementation Hospitals (RSPAD Gatot Soebroto Jakarta, RSUP Dr. Sardjito Yogyakarta and RSUP M. Djamil Padang) in the period 3 months after the issuance of Ethical Clearance and Approval for Implementation of Clinical Trials from BPOM.

The sample size is calculated using the following formula:

n1 = n2 = 2(Za+Z1-β)^2/ Δ^2

n1: the number of participants in the Exosome-MSC group n2: the number of participants in the control group Zα: standard deviation of type I error, 95% confidence interval (1.96) Zβ: standard deviation of type II error, power 80% (0.84) SD: standard deviation of duration of recovery on standard therapy (5.90). (Voinsky I, 2020)

Minimum expected difference in duration of healing (in days) when using Exosome-MSC compared to standard therapy (5) From the above calculation, the results of the calculation are N1 = N2 = 21.83 with rounding up each = 22 participants . To anticipate the adequacy of the number of participants , each group was added 8 participants , 30 participants each in the Exosome-MSC group and the control group so that the total number of participants was 60 participants.

Participants can be discontinued before the study is completed (drop-out) if they experience significant side effects and/or adverse events, both treatment related and non treatment related. Participants can also be discontinued before the study is completed (drop-out) if it worsens to a severe degree. All Participants will be discontinued from the study when the treatment and examination are completed according to the procedure.

Randomization of patients into the intervention group or control group was made for each study site through the block 4 randomization technique. This process will be coordinated by the Team who will carry out the Research Management/CRO function.

The double-blind procedure is a procedure to avoid bias of researchers and research participants that will affect the results of data analysis. To apply this procedure, the Exosome-MSC test material specimen in the Treatment Group was dissolved in 0.9% Nacl. The dosage form will be disguised so that it is similar to Nacl 0.9% in the Control Group. Research participants and local researchers implementing in hospitals do not have knowledge about the status of the research group (arm). During the study, patients continued to take their usual routine medications, such as antihypertensive drugs, antidiabetic drugs, calcium, or folic acid. The treatment will be included as a confounding factor.

Research participants will be monitored closely. CLINICAL examinations are carried out EVERY DAY, starting from the baseline (day 0) to day 14.

The clinical examination consists of:

1. body temperature,
2. oxygen saturation,
3. respiratory rate,
4. breath difficulties,
5. cough with phlegm,
6. RT-PCR results
7. standard therapy.received
8. allergic reactions,
9. secondary infection
10. side effects/ adverse events (AE) that are life threatening.
11. Remission score assessment based on 8 ordinal scales to determine Time to Clinical Improvement (TTCI).

TTCI is the number of days until clinical improvement can be observed, as indicated by a score of 1-3 out of 8 ordinal scales.

Laboratory examinations will be carried out on days 0, 1, 3, 7, 10 and 14 (unless they have been discharged/recovered first) . On days 0 and 7 when the Exosomes-MSC injection therapy is administered, laboratory examinations were performed before therapy.

Laboratory examinations consist of:

1. C-Reactive Protein,
2. ferritin,
3. D-Dimer,
4. LDH
5. Fibrinogen,
6. Routine blood, type count (including lymphocyte count)
7. PT and APTT
8. SGOT/SGPT,
9. urea/creatinine,
10. electrolyte K/Na/Cl,

Measures of intervention outcomes must be documented in a standardized Case Report Form (CRF) for each patient participating in the study.

Adverse Events are any events, whether predicted or not, which can be related to the test material or not, this includes worsening of the clinical condition previously owned by the participant.

Serious Adverse Events (SAE), include

1. Dead
2. Life threatening Inpatient / Participant requires treatment as an inpatient
3. Additional length of stay *
4. Permanent / significant disability
5. Congenital abnormalities

Additional length of stay, defined as length of stay at any time. Hospitalization due to routine administration of standard therapy is not included in this definition. If the participant experiences an adverse event during the hospitalization period, the condition must be reported as an adverse event.

All adverse events identified from the start of the study (day 0) to day 14 will be recorded in the adverse event form in the case report form (CRF).

In the event of a Serious Adverse Events (SAE), researchers at the research site must report it to Dermama Biotechnology Laboratorium within 24 hours after it is known as the initial report, the report is addressed to: Dr. dr. Indah Hidajati Kampono, Sp.DV(K) Dermama Biotechnology Laboratory Jl. Kelengkeng No. 8 Surakarta Phone/Fax Number: 0271-727007 E-mail: Indahhidajati01@gmail.com Telephone/Mobile Number: +62 811-2632-086

Written reports of serious adverse events must be sent to the Ethics Committee within 3 calendar days and to Indonesian National Agency of Food and Drugs Control (BPOM) within 7 calendar days for SAE that are fatal or life threatening, and within 15 calendar days for other SAE according to BPOM Regulation No. 21/201514.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with COVID-19 pneumonia confirmed by RT-PCR examination. Samples were obtained from nasopharyngeal swabs in patients with moderate
2. There is evidence of changes in chest X-ray with a picture of COVID-19 pneumonia and/or CT-Scan of the thorax with a ground glass opacity picture
3. Willing to participate in the study and sign the informed consent by the subject or family members.

Exclusion Criteria:

1. Diagnosed with mild COVID-19 pneumonia
2. Pregnant woman or positive pregnancy test
3. The subject is participating in another clinical trial.
4. Have a history of anaphylactic reactions, angioedema, or allergic reactions to antibiotics (penicillin and its derivatives) or other drugs.
5. Have an autoimmune disease
6. Have a history of malignancy
7. Undergoing hemodialysis or peritoneal dialysis
8. Recuring COVID-19 sufferers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to clinical improvement (days) | 14 days
  Clinical improvement is fulfilled with score 1-3 of the scale
  1. No hospitalization and no restrictions activity
  2. Not hospitalized, with activity restrictions, oxygen requirements at home, or both
  3. Hospitalized, does not require oxygen additional and no longer need maintenance ongoing medical treatment (used if hospitalization is extended for infection control or other reasons nonmedical)
  4. Hospitalized, not requiring supplemental oxygen but requiring ongoing medical care (related to COVID-19 or other medical conditions)
  5. hospitalized, requires supplemental oxygen
  6. hospitalized, requiring noninvasive ventilation or use high flow oxygen device;
  7. hospitalized, receiving mechanical ventilation invasive or extracorporeal membrane oxygenation (ECMO);
  8. deaths.

SECONDARY OUTCOMES:
Increase in Lymphocytes counts | 14 days
  Increase of Lymphocytes counts to normal range for adults between 1,000 and 4,800 x 10^3 per microliter of blood.
Decrease in D-dimer | 14 days
  Decrease of D-dimer from > 1000 ng/mL to normal range 220-500 ng/mL
Decrease in LDH level | 14 days
  Decrease in LDH level from > 300 U/L to normal range from 140 units per liter (U/L) to 280 U/L
Decrease in Ferritin concentration | 14 days
  Decrease in Ferritin concentration from > 500 ng/mL to below 300 ng/mL
Decrease in C-reactive protein | 14 days
  Decrease in C-reactive protein from > 10 mg/dL to normal range less than 10 mg/dL
Adverse events | 14 days
  Number of Adverse Events that occur during the study

CONTACTS AND LOCATIONS:
Overall Officials: Indah H Kampono, Dr. Sp.DV, Study Chair — Dermama; Bambang Darwono, Dr.Sp.OT, Principal Investigator — Research Center for Chemistry, National Research and Innovation Agency of Indonesia
Locations (3):
- Indonesia (3):
  - RSPAD Gatot Soebroto, Jakarta, DKI Jakarta
  - RSUP Dr. M. Jamil, Padang, West Sumatra
  - RSUP Dr. Sardjito, Yogyakarta

IPD SHARING:
Plan to Share IPD: No